CLINICAL TRIAL: NCT02465749
Title: Clinical Trials of Continuous Oxygen Therapy Combined With Blue Light Deprivation in the Treatment of Retinitis Pigmentosa
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Zhujiang Hospital (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou Jeeyor Medical Research Co.,Ltd. (Unknown)
Responsible Party: Principal Investigator, Qianying Gao, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZOC20150503
Record Dates: First submitted 2015-05-22; First posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; oxygen; blue light
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — Receptors, Antigen, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Continuous Oxygen (Experimental): Continuous oxygen intake and routine drug treatment .
  Interventions: Drug: Continuous oxygen; Drug: Compound thrombosis capsule sig: 1.5g/tid; Drug: Ginkgo biloba pills sig: 300mg/tid;; Drug: Vitamin B sig: 10mg/tid; Drug: Vitamin AD sig: 1 tablet/tid
- Blue Light Deprivation (Experimental): Wearing blue light-absorbing sunglasses at daily time and routine drug treatment
  Interventions: Device: blue light-absorbing sunglasses; Drug: Compound thrombosis capsule sig: 1.5g/tid; Drug: Ginkgo biloba pills sig: 300mg/tid;; Drug: Vitamin B sig: 10mg/tid; Drug: Vitamin AD sig: 1 tablet/tid
- Continuous Oxygen Therapy Combined With Blue Light Deprivation (Experimental): Continuous oxygen intake , Wearing blue light-absorbing sunglasses at daily time and routine drug treatment
  Interventions: Drug: Continuous oxygen; Device: blue light-absorbing sunglasses; Drug: Compound thrombosis capsule sig: 1.5g/tid; Drug: Ginkgo biloba pills sig: 300mg/tid;; Drug: Vitamin B sig: 10mg/tid; Drug: Vitamin AD sig: 1 tablet/tid
- control (Other): Routine drug treatment
  Interventions: Drug: Compound thrombosis capsule sig: 1.5g/tid; Drug: Ginkgo biloba pills sig: 300mg/tid;; Drug: Vitamin B sig: 10mg/tid; Drug: Vitamin AD sig: 1 tablet/tid

INTERVENTIONS:
Drug: Continuous oxygen — Continuous oxygen intake at a concentration of 93±3%, 3L/min flow-rate, 2h/bid, five days a week;
  Arms: Continuous Oxygen; Continuous Oxygen Therapy Combined With Blue Light Deprivation
Device: blue light-absorbing sunglasses — Wearing blue light-absorbing sunglasses at daily time;
  Arms: Blue Light Deprivation; Continuous Oxygen Therapy Combined With Blue Light Deprivation
Drug: Compound thrombosis capsule sig: 1.5g/tid — Compound thrombosis capsule sig: 1.5g/tid
Drug: Ginkgo biloba pills sig: 300mg/tid; — Ginkgo biloba pills sig: 300mg/tid;
Drug: Vitamin B sig: 10mg/tid — Vitamin B sig: 10mg/tid
Drug: Vitamin AD sig: 1 tablet/tid — Vitamin AD sig: 1 tablet/tid

SUMMARY:
The purpose of this study is to investigate the role of continuous oxygen therapy combined with blue light deprivation in prevention and control of retinitis pigmentosa, in order to find a new strategy of treatment for retinitis pigmentosa.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is one of of the major causes of blindness in ocular diseases.Up to now, the etiology of RP remained unclear, and there are no effective therapeutic methods. Several studies had showed that the retina of RP may be anoxic, and oxygen therapy, such as hyperbaric oxygen (hyperbaric oxygen, HBO) treatment, had shown a definite effect on RP. The investigators' previous researches also found that the retinal vessel oxygen saturation in patients with RP who were older than 40 years were significantly lower than normal controls, suggesting that oxygen may play an important role in the development of RP. Besides, many studies have revealed that blue light could damage retina pigment epithelium cells and photoreceptor cell specially. Therefore, investigators will combine continuous oxygen therapy and blue light deprivation therapy in the treatment for RP in this study, in order to find a new strategy of treatment for RP.

ELIGIBILITY:
Inclusion Criteria:

1. Severe patients with RP who meet the following criteria: (1) the EDTRS visual acuity of the good eye < 0.3 (low vision);(2) the radius of central visual field< 10 °(low vision)
2. Age range from 18 to 60 years old, sex unlimited
3. Able to adhere to treatment for more than 12 months
4. Willing to participate in this trial, and sign the informed consent

Exclusion Criteria:

1. Serious opacity of cornea, lens or vitreous body which can't have clear fundus examination
2. Patients with severe systemic diseases who was unable to tolerate the examinations, such as heart failure, respiratory failure, sepsis, severe anemia, kidney disease, history of eye surgery and so on
3. Patients who was unable to tolerate oxygen treatment, such as severe pulmonary edema, deformity of the respiratory tract, respiratory tract infection, tuberculosis, patients with pregnancy, and so on

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 404 (Estimated)
Dates: Start 2015-05; Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients preserved 80% of the initial visual acuity at 5 years follow-up. | at 5 years follow-up

SECONDARY OUTCOMES:
ERG b-wave mean values | at 5 years follow-up
Change of visual field | at 5 years follow-up
  visual field
Fundus changes of fluorescence fundus angiography | at 5 years follow-up
Retinal vessel oxygen saturation | at 5 years follow-up
  Retinal Oximetry
intra-ocular pressure | at 1, 2, 3, 4 and 5 years follow-up
blood pressure | at 1, 2, 3, 4 and 5 years follow-up
Finger pulse oxygen saturation | at 1, 2, 3, 4 and 5 years follow-up
  Finger pulse oximetry
the mutant genes of retinitis pigmentosa | at admission
  gene screening

CONTACTS AND LOCATIONS:
Overall Officials: Qianying Gao, PHD, Principal Investigator — State Key Laboratory of Ophthalmology,Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- State Key Laboratory of Ophthalmology,Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China